CLINICAL TRIAL: NCT00152893
Title: The Effects of Chromium Supplementation on Glucose and Lipid Metabolism in Patients With HIV Infection
Brief Title: To Determine if Chromium Nicotinate Supplementation Will Improve Insulin Resistance in HIV Patients With Metabolic Abnormalities
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johane Allard (Other)
Collaborators: Canadian Foundation for AIDS Research (CANFAR) (Other)
Responsible Party: Sponsor-Investigator, Johane Allard, Gastroenterologist, Prof. of Medicine, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 03-0703-A; 015 027
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections
Keywords: HIV; blood sugar > 6.1 mmol/l; triglycerides > 2 mmol/l; total cholesterol > 5.5 mmol/l or HDL < 0.9 mmol/l
MeSH Terms: conditions — HIV Infections | interventions — chromium nicotinic acid complex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Chromium (Experimental): 400 μg (200 μg pills, twice per day) of Cr-nicotinate
  Interventions: Drug: chromium nicotinate
- Placebo (Placebo Comparator): Identical looking placebo (di-calcium phosphate)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: chromium nicotinate
  Arms: Chromium
Drug: Placebo
  Arms: Placebo

SUMMARY:
In HIV patients, fasting insulin levels decrease with chromium supplementation. This study is to determine if chromium nicotinate supplementation at 400ug/day for 16 weeks will improve insulin resistance in HIV patients with metabolic abnormalities.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, crossover study where patients will be supplemented for 16 weeks with either chromium nicotinate 400 ug/day or placebo and then crossover to the opposite treatment for another 16 weeks. Each soft gel capsule of chromium contains 200ug of chromium and patients will take 1 capsule twice a day or its placebo. Placebo contains di-calcium phosphate in a soft gel capsule and its appearance is similar to the chromium capsules.

ELIGIBILITY:
Inclusion Criteria:

* HIV documented patients will be considered for the study if they have at least one abnormality with respect to fasting blood glucose, TG, total or HDL cholesterol. Normal fasting glucose is defined as < 6.1 mmol/L. Hypertriglyceridemia is defined as concentrations above 2.0 mmol/L on the basis of reports of increased risk of cardiac disease. Hypercholesterolemia is defined as concentrations above 5.5 mmol/L and a low HDL-cholesterol concentration as less than 0.9 mmol/L.
* Patients will need to be on a stable drug regimen for at least 8 weeks and not taking any chromium supplement or chromium-containing multivitamins 4 weeks prior to and during the study period. Patients can stay on their hypoglycemic or lipid-lowering medications and the required dosage will be monitored.

Exclusion Criteria:

* Patients will be excluded if there is concomitant acute infection or malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2002-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
insulin resistance calculated using fasting glucose and fasting insulin levels in blood | BL & 16 weeks
  HOMA-IR

SECONDARY OUTCOMES:
hemoglobin A1c (HbA1c) | BL & 16 weeks
blood lipid profile (triglycerides [TG], cholesterol or high-density lipoprotein [HDL]) | BL & 16 weeks
body composition by dual energy x-ray absorptiometry (DEXA) scan, bioelectric impedance analysis and skin fold measurement | BL & 16 weeks
oxidative stress | BL & 16 weeks
plasma chromium | BL & 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johane Allard, MD, FRCPC, Principal Investigator — University Health Network - Toronto General Hospital
Locations (1):
- University Health Network - Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Aghdassi E, Arendt B, Salit IE, Allard JP. Estimation of body fat mass using dual-energy x-ray absorptiometry, bioelectric impedance analysis, and anthropometry in HIV-positive male subjects receiving highly active antiretroviral therapy. JPEN J Parenter Enteral Nutr. 2007 Mar-Apr;31(2):135-41. doi: 10.1177/0148607107031002135. PMID 17308254
- [Result] Aghdassi E, Arendt BM, Salit IE, Mohammed SS, Jalali P, Bondar H, Allard JP. In patients with HIV-infection, chromium supplementation improves insulin resistance and other metabolic abnormalities: a randomized, double-blind, placebo controlled trial. Curr HIV Res. 2010 Mar;8(2):113-20. doi: 10.2174/157016210790442687. PMID 20163347
- [Result] Arendt BM, Aghdassi E, Mohammed SS, Fung LY, Jalali P, Salit IE, Allard JP. Dietary intake and physical activity in a Canadian population sample of male patients with HIV infection and metabolic abnormalities. Curr HIV Res. 2008 Jan;6(1):82-90. doi: 10.2174/157016208783571973. PMID 18288980